CLINICAL TRIAL: NCT00944749
Title: Horse ATG/CsA in Aplastic Anemia Patients Unresponsive to or With a Suboptimal Response to Rabbit ATG/CsA Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090183; 09-H-0183
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-09

CONDITIONS: Anemia, Aplastic; Anemia, Hypoplastic
Keywords: H- ATG; Anti -Thymocyte Globulin; Lymphocyte Immune Globulin; Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Antilymphocyte Serum; Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: h-ATG (ATGAM ); Drug: Cyclosporine (Gengraf )

INTERVENTIONS:
Drug: h-ATG (ATGAM )
Drug: Cyclosporine (Gengraf )

SUMMARY:
Background:

* Severe plastic anemia can lead to problems with bone marrow platelet production and result in low blood platelet counts, which require frequent platelet transfusions to improve blood clotting.
* A standard treatment for SAA involves injections of rabbit-antithymocyte globulin (r-ATG). r-ATG is developed by injecting horses with a type of human white blood cells called thymocytes. The horse's immune system reacts against these cells and makes antibodies that can destroy them. These antibodies are collected and purified to make r-ATG. Horses can also be used for this procedure to make horse-antithymocyte globulin (h-ATG).
* h-ATG is approved by the Food and Drug Administration for the treatment of aplastic anemia. h-ATG is a standard first-line method to treat aplastic anemia, but researchers do not know how effective it is in patients who were first treated unsuccessfully with r-ATG.

Objectives:

- To evaluate the effectiveness and safety of horse-ATG (with cyclosporine) in increasing blood counts and reducing the need for transfusions in aplastic anemia patients who have failed to respond to prior immunosuppressive treatment with rabbit-ATG and cyclosporine.

Eligibility:

- Patients 2 years of age and older who have consistently low blood platelet counts related to aplastic anemia that has not responded to conventional treatment with rabbit-ATG.

Design:

* After initial screening, medical history, and blood tests, patients will be admitted to the inpatient unit at the National Institutes of Health Clinical Center. Researchers will perform a skin test with h-ATG to check for allergic or other adverse reaction.
* After the skin test, h-ATG will be given into a vein continuously over 4 days.
* Cyclosporine will also be given to improve the response rate of ATG treatment. Treatment with cyclosporine will start the same day as the h-ATG, either in liquid or capsule form, and continued for 6 months. The dose of cyclosporine will be monitored and adjusted based on blood levels and signs of side effects in the kidney and liver.
* To prevent or treat infections that may result from cyclosporine s effect on the immune system, patients will also take inhaled or capsule doses of pentamidine.
* After the study is completed, patients will have followup evaluations every 3 months, 6 months, and annually for 5 years. Evaluations will include blood samples and periodic bone marrow biopsies.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA), characterized by pancytopenia and a hypocellular bone marrow, is effectively treated by immunosuppressive therapy, usually a combination of antithymocyte globulin (ATG) and cyclosporine (CsA). Survival rates following this regimen are equivalent to those achieved with allogeneic stem cells transplantation. However, approximately 1/3 of patients will not show blood count improvement after ATG/CsA. General experience and small pilot studies have suggested that such patients benefit from further immunosuppression. Furthermore, analysis of our own clinical data suggests that patients with minimal blood count responses to a single course of ATG, even when transfusion independence is achieved, have a markedly worse prognosis than patients with robust hematologic improvement.

The majority of the experience in the US and worldwide has been with horse ATG (h-ATG) plus CsA as initial therapy in SAA. Rabbit ATG (r-ATG) plus CsA has been employed successfully in about 1/3 of cases in those who are refractory to initial h-ATG/CsA (current NHLBI Protocol 03-H-0249). In recent years, h-ATG and r-ATG have been used interchangeably in treatment-naive patients, and initial therapy with r-ATG/CsA is now frequent in the US and the only option in Europe and Japan, where h-ATG is no longer available. An active NHLBI randomized study is comparing the efficacy of h- and r-ATG as initial therapy in SAA, and the results from a recently completed interim analysis suggest that the hematologic response rate ultimately may not be comparable between these two agents (Protocol 06-H-0034). There is no published report on the outcome of repeat immunosuppressive therapy in those patients refractory to initial r-ATG/CsA, and thus the management of these patients is uncertain. We therefore propose this study of h-ATG/CsA in SAA patients who are refractory or have a suboptimal response to r-ATG.

The primary endpoint will be the response rate at 3 months where response is defined as no longer meeting criteria for SAA.

The primary objective is to evaluate the effectiveness (response rate) at 3 months of a second course of immunosuppression with h-ATG/CsA in subjects refractory to or with a suboptimal response to a course of r-ATG/CsA or cyclophosphamide at least 3 months post treatment.

Secondary objectives include robustness of hematologic recovery, relapse, response rate at 6 months, clonal evolution and overall survival.

The primary endpoint will be changes in absolute neutrophil count, platelet count, reticulocyte count at 3 months.

Secondary endpoints will include time to relapse, changes in cytogenetics, time to death.

ELIGIBILITY:
* All patients 2 years old or over with SAA who have failed initial immunosuppression with r-ATG/CsA and are not candidates for a matched sibling marrow transplantation will be considered for enrollment. Patients who have a suitable matched sibling donor will be referred for consideration of allogeneic bone marrow transplantation. Patients not willing to undergo transplantation will be considered for enrollment. Eligibility will be determined on another screening Hematology Branch protocol (97-H-0041) or another active Hematology branch protocol. The time between determination of eligibility and signing consent to participate on this protocol and initiate treatment on this protocol will not exceed 90 days.

INCLUSION CRITERIA:

1. Diagnosed with SAA characterized by:

   1. Bone marrow cellularity < 30% (excluding lymphocytes)
   2. At least two of the following:

   i. Absolute neutrophil count <500/ microL

   ii. Platelet count <20,000/ microL

   iii. Reticulocyte count <60,000/ microL
2. Failure to respond to an initial course of r-ATG/CsA or cyclophosphamide at least 3 months post-treatment or a suboptimal response to initial therapy defined by both platelet and reticulocyte count < 50,000 /microL at 3 months post-treatment
3. Age greater than or equal to 2 years of age

EXCLUSION CRITERIA:

1. Diagnosis of Fanconi anemia. Patients with very severe neutropenia (ANC < 200 /microL) will not be excluded initially if results of Fanconi anemia testing are not available or pending. If evidence of Fanconi anemia is later identified, the subject will go off study.
2. Evidence of a clonal disorder on cytogenetics. Patients with very severe neutropenia (ANC < 200/uL) will not be excluded initially if results of cytogenetics are not available or pending. If evidence of a clonal disorder is later identified, the subject will go off study.
3. Patients who received prior course(s) of alemtuzumab will not be excluded.
4. Infection not adequately responding to appropriate therapy
5. HIV seropositivity
6. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy or that death within 7-10 days is likely.
7. Subjects with cancer who are on active chemotherapeutic treatment or who take drugs with hematological effects will not be eligible
8. Serum creatinine > 2.5 mg/dL
9. Current pregnancy, breast-feeding or unwillingness to refrain from pregnancy if of child bearing potential
10. Inability to understand the investigational nature of the study or give informed consent

Ages: 2 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08-31 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Townsley, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mendez G Jr, Russell E. Gastrointestinal varices: percutaneous transheptic therapeutic embolization in 54 patients. AJR Am J Roentgenol. 1980 Nov;135(5):1045-50. doi: 10.2214/ajr.135.5.1045. PMID 6778145
- [Background] Maciejewski JP, Selleri C, Sato T, Anderson S, Young NS. Increased expression of Fas antigen on bone marrow CD34+ cells of patients with aplastic anaemia. Br J Haematol. 1995 Sep;91(1):245-52. doi: 10.1111/j.1365-2141.1995.tb05277.x. PMID 7577642
- [Background] Risitano AM, Maciejewski JP, Green S, Plasilova M, Zeng W, Young NS. In-vivo dominant immune responses in aplastic anaemia: molecular tracking of putatively pathogenetic T-cell clones by TCR beta-CDR3 sequencing. Lancet. 2004 Jul 24-30;364(9431):355-64. doi: 10.1016/S0140-6736(04)16724-X. PMID 15276395
- [Derived] Zaimoku Y, Patel BA, Adams SD, Shalhoub R, Groarke EM, Lee AAC, Kajigaya S, Feng X, Rios OJ, Eager H, Alemu L, Quinones Raffo D, Wu CO, Flegel WA, Young NS. HLA associations, somatic loss of HLA expression, and clinical outcomes in immune aplastic anemia. Blood. 2021 Dec 30;138(26):2799-2809. doi: 10.1182/blood.2021012895. PMID 34724566
- [Derived] Scheinberg P, Townsley D, Dumitriu B, Scheinberg P, Weinstein B, Rios O, Wu CO, Young NS. Horse antithymocyte globulin as salvage therapy after rabbit antithymocyte globulin for severe aplastic anemia. Am J Hematol. 2014 May;89(5):467-9. doi: 10.1002/ajh.23669. Epub 2014 Mar 7. PMID 24415649
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0183.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Subjects were given a second course of immunosuppression with h-ATG/CsA in subjects' refractory to or with a suboptimal response to a course of r-ATG/CsA or cyclophosphamide at least 3 months post-treatment
Period: Overall Study
Arm/Group | Single Arm
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 16
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 7
  More than one race | 1
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response at 3 Months.
Description: The primary endpoint was hematologic response at 3 months, defined as no longer meeting criteria for Severe Aplastic Anemia (SAA) defined as bone marrow cellularity of less than 30% and severe pancytopenia with at least two of the following peripheral blood count criteria: (i) absolute neutrophil count less than 0.5×109/L; (ii) absolute reticulocyte count less than 60×109/L; and (iii) platelet count less than 20×109/L.
  A complete response was defined as absolute neutrophil count (ANC) above 1.0×109/L, Hgb > 10 g/dL, and platelet count > 100×109/L.
  A partial response was defined as a hematologic response that was not sufficient for a complete response.
Time Frame: 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 22
Participants | 0

2. Primary Outcome: Number of Participants With Complete Response at 3 Months.
Description: The primary endpoint was hematologic response at 3 months, defined as no longer meeting criteria for Severe Aplastic Anemia (SAA).
  A complete response was defined as absolute neutrophil count (ANC) above 1.0×109/L, Hgb > 10 g/dL, and platelet count > 100×109/L.
  A partial response was defined as a hematologic response that was not sufficient for a complete response.
  In subjects with a non-robust hematologic response at 3 months, improvement in one or more of the listed peripheral blood parameter (a,b,c) were recorded as a response: a) ANC - if baseline ANC below 0.5×109/L, increase in ANC by > 0.3×109/L, if baseline ANC above 0.5×109/L, any increase in ANC by > 0.5×109/L of blood; (b) platelets - if baseline platelet count < 50×109/L, any increase in platelet count by > 20×109/L of blood; c) hemoglobin - any increase in hemoglobin by 1.5 g/dl of blood in transfusion-independent patients and in absolute reticulocyte count to > 60×109/L of blood in transfusion-dependent patients.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 22
Participants | 2

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 14/23
Other Adverse Events (participants affected / at risk) | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=23)
Hospitalization - Neutropenic fever (Blood and lymphatic system disorders) | 7
Hospitalization - Infection/ Febrile neutropenia (Infections and infestations) | 2
Hospitalization - Hemorrhage/ bleeding (Blood and lymphatic system disorders) | 1
Death - Hemorrhage/ bleeding (Blood and lymphatic system disorders) | 1
Hospitalization - Infection (Infections and infestations) | 9
Hospitalization - Gastrointestinal (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=23)
Rhinorrhea (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes